CLINICAL TRIAL: NCT07287696
Title: Effect of Siwan Sand Therapy on Pulmonary Functions of Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Nashwa Mohammed Alaa Allam, lecturer, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC\012\001198
Record Dates: First submitted 2025-05-19; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: siwa,traditional therapy ,rheumatoid arthritis,pulmonary function
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: a prospective, randomized, single blind, pre and post-test, clinical trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: sand therapy — Patients received sand bathing between 2 pm and 4 pm between the end of May and the first two weeks of September. The atmospheric temperature was 40-45°C, the sand surface temperature ranged from 75 to 82°C and the temperature under the sand surface by 10-20 cm was 50-60°C, measured by an infrared thermometer (Medisana, Germany).
  A hole of 20-40 cm in depth, 80 cm in width and 100-150 cm in length was dug. A long shallow hole was dug in the early morning to permit the heating of the sand by the sun's rays; after the lying down the patient, he/she was covered to the neck by hot dry sand from the surface of the desert.
Other: physical therapy program — physical therapy program composed of aerobic and strengthening exercise, TENS and hot application 2 sessions per week for 2 months. Group (B): consisted of 15 patients who were treated by the Siwan traditional program consisting of 5-sessions of sand therapy for 5 days followed by massage with olive oil.
  Physiotherapy Aerobic exercises in the form of walking on a treadmill, with moderate intensity ranged from 55-65% of target heart rate, according to Karvonen formula {resting heart rate + (maximum heart rate - resting hart rate)55-65%}[33]; the patient performed intermittent aerobic exercise for 15-30 min at the first session; they began with 15 min walking and then the duration was increased to reach 30 min; patients began with warming up for 5-minutes, followed by stimulus phase for 5-20 minutes and ended with cooling down for 5-minutes. The patient performed walking as a home program for Two times per week. Moreover, the physiotherapy program involved progressive strengthen

SUMMARY:
The purpose of this study was to compare between the effects of Siwan sand therapy and physical therapy program on pulmonary function, functional activity, and pain in rheumatoid arthritis patients.

Forty five patients were recruited according to the American Rheumatism Association criteria 2010 for the study, fifteen of them had been dropped, the other thirty patients (11 male and 19 female) were assigned into two equal groups: group (A) received Siwan sand therapy inform of sand bath for 5-days, followed by massage with olive oil, while group (B) received physiotherapy for 2-months in form of hot back, TENS, aerobic exercise and strengthening exercise, for the period between June 2016 and August 2019. All patients were evaluated pre-treatment and post treatment

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized, single blind, pre and post-test, clinical trial. Approval of the Ethical Committee was obtained from the institutional review board at Faculty of physical therapy, Cairo University before study started. The study was followed the Guidelines of Declaration of Helsinki on the conduct of human research. The study was conducted for the period between June 2016 and August 2019.

Study participants A sample of forty five RA patients, from both gender. from Ekasr Eleiny hospital, and from other private clinic located in Cairo were recruited to participate in the study. They were interviewed individually to assess their eligibility to be included in the study. They were assessed and treated at Cairo University out patients clinic, private clinic and in Siwa oasis traditional healing center in Marsa Matrouh Governorate, pre and post pulmonary function test performed in fitness and rehabilitation unite in Elaser Elainy hospital.

The inclusion criteria were definite RA that fulfilled the 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for RA [31], Patients were on their stable doses of anti-rheumatic drugs, Patients with moderate, severe rheumatoid arthritis, they had positive RF and anti-CCP, Both sexes participated in this study, their ages range from 25 to 59 years, body mass index from 25 to 30, Pain of at least 3 mm on a visual analogue scale (VAS) from 0 mm (no pain) to 10 mm (worst imaginable pain), Patients with (I) complete functional capacity with ability to carry out all usual duties without handicaps, (II) functional capacity adequate to conduct normal activities despite handicap of discomfort or limited mobility of one or more joints, (III) functional capacity adequate to perform only a few or none of the duties of usual occupation or of self-care [16].

Patients who were known to have one of the following criteria were excluded from the study: uncontrolled arterial hypertension [systolic blood pressure (SBP) ≥ 180 mm Hg and/or diastolic blood pressure (DBP) ≥ 100 mm Hg] 32 (Tanaka and Kazumi, 1990). Uncontrolled diabetes, Previous renal transplanted patients, Patients had coronary artery disease including: unstable angina, Pregnant woman's, Bleeding disorder, Largely or wholly incapacitated with patient bedridden or wheel chair bound, permitting little or no self-care.

Randomization Fifteen patients had been dropped, two of them were misdiagnosed, one of them have disc prolapse that prevent here from traveling from Cairo to Siwa as it was a long distance, some of them refused to complete the physical therapy sessions as they felt that there was not any improvement in their cases, one of them had had depression and anxiety she refused to complete the sessions, some of them refused to perform pulmonary function test after sessions as they were afraid of transmission of infection. The other 30 (11 male and 19 female) patients were randomly assigned into two groups by a blinded and an independent research assistant who opened sealed envelopes that contained a computer generated randomization card. Written informed consent was obtained from all participants before the baseline evaluation.

Intervention Group (A): consists of 15 patients who were treated by the physical therapy program composed of aerobic and strengthening exercise, TENS and hot application 2 sessions per week for 2 months. Group (B): consisted of 15 patients who were treated by the Siwan traditional program consisting of 5-sessions of sand therapy for 5 days followed by massage with olive oil.

Physiotherapy Aerobic exercises in the form of walking on a treadmill, with moderate intensity ranged from 55-65% of target heart rate, according to Karvonen formula {resting heart rate + (maximum heart rate - resting hart rate)55-65%}[33]; the patient performed intermittent aerobic exercise for 15-30 min at the first session; they began with 15 min walking and then the duration was increased to reach 30 min; patients began with warming up for 5-minutes, followed by stimulus phase for 5-20 minutes and ended with cooling down for 5-minutes. The patient performed walking as a home program for Two times per week. Moreover, the physiotherapy program involved progressive strengthening exercises for lower extremity, to strength flexor, extensor, adductor, abductor, internal and external rotator of hip joint, also flexor and extensor of knee joint, and ankle dorsi flexors. The patients also performed upper extremity strengthening exercise for shoulder flexor extensor, and abductors, also strengthening of elbow flexors and extensors, wrist flexors and extensor were performed.

The positions of patients differ according to the muscle group that should be strengthen, so the positions were sitting, supine or standing side lying position. Frequency of exercise was two time per week for two months. Isometric exercises provided sufficient muscle tone with no aggravation of clinical disease activity in case of acutely inflamed joints. Moderate contraction was held for 5-10 seconds, 5-20 repetitions, 3 set. However, in case of low disease activity, exercises were performed using very low weights 30% of one repetition max.

Heat used before exercise for maximum benefit [34]. Patient in relaxed position, the hot pack wrapped by 2 layer of towel and applied on the affected joints especially for about 20 minutes.

ATranscutaneous Electrical Nerve Stimulation (TENS): using Burst-mode, in burst mode the carrier frequency of the current is high (70-100 Hz), but it is delivered in small bursts at a low rate (3-4 bursts per second). Electrode placements are placed on the painful joints.

Siwan traditional therapy Fifteen patients received Siwan traditional therapy in the form of sand bathing, and massage with olive oil every day for 5 days. Patients received sand bathing between 2 pm and 4 pm between the end of May and the first two weeks of September. The atmospheric temperature was 40-45°C, the sand surface temperature ranged from 75 to 82°C and the temperature under the sand surface by 10-20 cm was 50-60°C, measured by an infrared thermometer (Medisana, Germany).

A hole of 20-40 cm in depth, 80 cm in width and 100-150 cm in length was dug. A long shallow hole was dug in the early morning to permit the heating of the sand by the sun's rays; after the lying down the patient, he/she was covered to the neck by hot dry sand from the surface of the desert.

Before sand bathing patients were advised not to take a shower or to use body lotion or cream during the sand bathing period and for three days after treatment, they were not permitted to use fan or air conditioning, they should cover their bodies well as to prevent air draft and drink lots of hot or warm fluids before and after every session (e.g. anise and lemon juice).

The burial lasted approximately 20 min. Once the sand became wet with sweat, it was replaced by fresh hot sand. Next, the patient was wrapped in a towel and remained for 15 min in a well-sealed tent pitched near the burial area. Patients drank liquids like anise and lemon juice to avoid dehydration; drinking water was forbidden at this point. Patients were wrapped to avoid wind or air draft, which might have negative consequences (e.g. muscle stiffness or pounding).

The body returned to the normal temperature and regained its resting status during the time spent in the tent. Then, patients were allowed to go to the hotel, rested in their beds; sweating continued two hours post session; after the sweating stopped, they were allowed to change their clothes with dry ones.

Outcome measures

Pulmonary function:

Measured by spirometer, pulmonary function test performed for both group before and immediately after intervention, FVC was measured by asking the patient to take deep inspiration and then forcefully expire the air in the mouth piece of spirometer as fast as he could. FEV1 volume of air measured in the first second of forced expiration.

B. Functional disability:

Measured by functional disability questionnaire, the patients were asked the questions of disability before and after intervention. By interviewing the patients personally and asking them the questions in the questionnaire.

C. pain severity:

It was measured by Visual analog scale (VAS) every patient in both group was asked to choose a number from 1 to 10 that represent his feeling of pain, before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were definite RA that fulfilled the 2010 American College of Rheumatology/European League Against Rheumatism classification criteria for RA

* Patients were on their stable doses of anti-rheumatic drugs
* Patients with moderate, severe rheumatoid arthritis
* they had positive RF and anti-CCP
* Both sexes participated in this study
* their ages range from 25 to 59 years
* body mass index from 25 to 30
* Pain of at least 3 mm on a visual analogue scale (VAS) from 0 mm (no pain) to 10 mm (worst imaginable pain)
* Patients with (I) complete functional capacity with ability to carry out all usual duties without handicaps, (II) functional capacity adequate to conduct normal activities despite handicap of discomfort or limited mobility of one or more joints, (III) functional capacity adequate to perform only a few or none of the duties of usual occupation or of self-care -

Exclusion Criteria:

* uncontrolled arterial hypertension [systolic blood pressure (SBP) ≥ 180 mm Hg and/or diastolic blood pressure (DBP) ≥ 100 mm Hg] 32 (Tanaka and Kazumi, 1990).
* Uncontrolled diabetes,
* Previous renal transplanted patients,
* Patients had coronary artery disease including: unstable angina,
* Pregnant woman's,
* Bleeding disorder,
* Largely or wholly incapacitated with patient bedridden or wheel chair bound, permitting little or no self-care.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 2 year
  Measured by spirometer, pulmonary function test performed for both group before and immediately after intervention, FVC was measured by asking the patient to take deep inspiration and then forcefully expire the air in the mouth piece of spirometer as fast as he could. FEV1 volume of air measured in the first second of forced expiration.

SECONDARY OUTCOMES:
Functional disability | 2 year
  Measured by functional disability questionnaire, the patients were asked the questions of disability before and after intervention. By interviewing the patients personally and asking them the questions in the questionnaire
pain severity | 2 year
  It was measured by Visual analog scale (VAS) every patient in both group was asked to choose a number from 1 to 10 that represent his feeling of pain, before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Egypt